CLINICAL TRIAL: NCT03432546
Title: Acute and Persistent Pain in Intensive Care Patients
Brief Title: Acute and Persistent Pain in ICU Patients
Acronym: PAIN-ICU
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Töölö Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HUS/2779/2017
Record Dates: First submitted 2017-12-20; First posted 2018-02-14 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Critical Care; Acute Pain; Chronic Pain
MeSH Terms: conditions — Acute Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients: Over 18-year old intensive care patients, non-interventional prospective observational study
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Non-interventional

SUMMARY:
Approximately 20,000 patients are treated in intensive care units (ICU) in Finland annually. During ICU stay many diagnostic and other procedures as well as immobilization and underlying diseases may cause pain. Therefore the incidence of pain in ICU patients can be high. Acute pain may cause several detrimental effects including respiratory distress, tissue hypoxia, immunosuppression and anxiety. After discharge many survivors of critical care have lower health-related quality of life, symptoms of post-traumatic stress disorder or persistent pain.

Only few studies with a focus on acute or persistent pain in ICU patients have been made, hence the incidence and risk factors for ICU-related pain is not very well known. Some of the identified risk factors for persisting pain may be increased age, sepsis or inadequate pain management during ICU stay. Opioids are most often used for analgesics in intensive care. Because they may have several adverse effects the use must be based on validated pain scales. Many factors such as sedation, relaxation or delirium of the patient complicates the management of the pain.

This prospective observational study aims to determine the incidence and risk factors for acute and persistent pain in ICU patients as well as and the use of analgesics during intensive care.

DETAILED DESCRIPTION:
This prospective observational study aims to determine the incidence and risk factors for acute and persistent pain in ICU patients as well as and the use of analgesics during intensive care.

The recruitement process is finished, but the follow-up is on-going. Patients are followed-up by subsequent questionnaires until 5 years after admission to the ICU.

ELIGIBILITY:
Inclusion Criteria:

* not meeting the exclusion criteria

Exclusion Criteria:

* pregnant patients
* age under 18 years
* suffering from significant brain injury
* elective neurosurgical patients
* probable organ donors
* suffering from significant cognitive impairment
* presumed death under 48h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective cohort of intensive care patients
Sampling Method: Non-Probability Sample
Enrollment: 707 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of acute pain | Through study completion, an average of 3 days
  Moderate or severe pain (numerical rating scale (NRS) value above 3 / critical pain observatory tool (CPOT) value ≥3) during intensive care
Incidence of persistent neuropathic pain using Pain Detect | At intensive care follow up clinic at three months after discharge and thereafter the change in pain annually for 5 years
  Moderate or severe pain.
Incidence of anxiety affecting persistent pain | At intensive care follow up clinic at three months after discharge and thereafter the change in anxiety annually for 5 years
  State Trait anxiety Index T (STAI-T)

SECONDARY OUTCOMES:
Analgesic use | Through study completion, an average of 3 days
  Analgesics administered during intensive care including indications and dosages
Delirium | Through study completion, an average of 3 days
  Incidence of delirium during intensive care by using Intensive Care Delirium Screening Checklist (ICDSC, scores 0-8) scale, a sum of symptoms equal or above 4 is considered affirmative for delirium

CONTACTS AND LOCATIONS:
Overall Officials: Maija-Liisa Kalliomäki, Study Chair — Tampere University Hospital; Otto Mäkinen, Study Chair — Tampere University; Sari Karlsson, Study Chair — Tampere University Hospital; Simo Varila, Study Chair — Tampere University Hospital; Minna Peltomaa, Study Chair — Tampere University Hospital; Karita Koskinen, Study Chair — HUS; Anna-Maria Kuivalainen, Study Chair — HUS; Katri Hamunen, Study Chair — HUS Pain Clinic; Minna Bäcklund, Study Chair — HUS; Sari Sutinen, Study Chair — HUS; Leena Pettilä, Study Chair — HUS; Annika Laukkanen, Study Chair — Töölö Hospital
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Meilahti, Helsinki
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: No